CLINICAL TRIAL: NCT00974935
Title: Phase I Study of the Safety and Immunogenicity of Recombinant Staphylococcal Enterotoxin B Vaccine (STEBVax) in Healthy Adults
Brief Title: Phase I STEBVax in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0009; HHSN272200800006C
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2014-09

CONDITIONS: Toxic Shock Syndrome Staphylococcal
Keywords: Staphylococcal enterotoxin B, vaccine, Staphylococcus aureus, toxic shock syndrome
MeSH Terms: conditions — Staphylococcal Infections; Shock, Septic | interventions — Aluminum Hydroxide

ARMS (7):
- Cohort 1 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 0.01 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 2 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 0.1 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 3 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 0.5 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 4 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 2.5 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 5 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 10 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 6 (Experimental): Single dose of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 20 mcg intramuscular.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine
- Cohort 7 (Experimental): Two doses of staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 20 mcg intramuscular 21 days apart.
  Interventions: Drug: Aluminum hydroxide; Biological: STEBVax vaccine

INTERVENTIONS:
Drug: Aluminum hydroxide — Single dose of recombinant staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 0.01, 0.1, 0.5, 2.5, 10 or 20 mcg intramuscular and 2 doses of 20 mcg intramuscular 21 days apart. STEBVax vaccine will be administered as a single 0.5 mL intramuscular injection into the deltoid muscle of the non-dominant arm; subjects in the 2 dose cohort will have the vaccine administered in the alternate arm.
Biological: STEBVax vaccine — Single dose of recombinant staphylococcal enterotoxin B vaccine (STEBVax) in Alhydrogel adjuvant at 0.01, 0.1, 0.5, 2.5, 10 or 20 mcg intramuscular and 2 doses of 20 mcg intramuscular 21 days apart. STEBVax vaccine will be administered as a single 0.5 mL intramuscular injection into the deltoid muscle of the non-dominant arm; subjects in the 2 dose cohort will have the vaccine administered in the alternate arm.

SUMMARY:
The main purpose of this study is to test the safety of a new vaccine, STEBVax, which may lead to a useful treatment for toxic shock syndrome. The second purpose is to determine whether STEBVax causes the body to produce antibodies (proteins that fight infection) to help the body resist disease. Researchers expect STEBVax shots will cause the development of antibodies in the blood. Study participants will include up to 42 healthy adults, ages 18-40, from the University of Maryland Baltimore community. Participants will be assigned to one of 7 vaccine dose groups. Assignment to dosage groups will depend on when individuals are enrolled in the study. Study procedures will include blood sampling, urine collection, and physical examinations. Subjects will maintain a memory aid documenting daily oral temperatures and possible vaccine side effects. Participants will be involved in study related procedures for up to 201 days.

DETAILED DESCRIPTION:
This study is a Phase I study of the safety and immunogenicity of recombinant Staphylococcal Enterotoxin B vaccine (STEBVax) in healthy adults. STEBVax is a recombinant mutated form of staphylococcal enterotoxin B (SEB) containing three point mutations that disrupt the interaction of the toxin with human major histocompatibility complex (MHC) class II receptors and render the protein non-toxic while retaining most of the immunogenicity. The primary intended result of this program is the development of a hyperimmune serum for treatment of toxic shock syndrome (TSS) originating from nosocomial, environmental or potential bioterrorist events. An additional long-term goal is the development of a multivalent vaccine and immunotherapeutic for treating or preventing diseases caused by Staphylococcus (S.) aureus. The long-range goal is to develop a vaccine that will protect against a broad range of staphylococcal superantigens. The primary objective is to evaluate and assess the safety of parenterally administered STEBVax vaccine in healthy adult subjects over a range of doses from 0.01 to 20 mcg by intramuscular injection. The secondary objectives are to determine the immunogenicity of STEBVax vaccine over a range of doses as determined by the rate and titer of seroconversion with serum anti-S. aureus enterotoxin B IgG antibodies measured by enzyme-linked-immunosorbent serologic assay (ELISA). Participants will include 28 healthy adult subjects from the University of Maryland Baltimore community. Subjects will receive a dose of STEBVax in Alhydrogel adjuvant at one of the following doses: 0.01, 0.1, 0.5, 2.5, 10 or 20 mcg or 2 doses of 20 mcg given 21 days apart. STEBVax will be administered as a single 0.5 mL intramuscular injection. Subjects will be followed for safety, reactogenicity, and immune response after vaccination. Subjects will be observed in the clinic for at least 8 hours after vaccination and remain in the Baltimore-Washington metropolitan area for 7 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Age 18 - 40 years, inclusive.
* Good "general health" as determined by vital signs (heart rate <100 bpm; blood pressure systolic > 90 mm Hg and less than or equal to 140 mm Hg; diastolic > 50 mm Hg and less than or equal to 90 mm Hg; oral temperature <100.4 degrees Fahrenheit), medical history, and a physical examination within 45 days before administration of Recombinant Staphylococcal Enterotoxin B Vaccine (STEBVax). Blood pressure outside this range may be repeated once on another occasion.
* Expressed interest and availability to fulfill the study requirements
* Agrees not to become pregnant from the time of study enrollment until at least 90 days after the last administration of STEBVax; if a woman is sexually active and capable of conception (i.e., no history of hysterectomy or tubal ligation), she must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), condoms with spermicidal agents, or must have a vasectomized partner, or must be sexually abstinent. A woman is eligible if she is monogamous with a vasectomized male
* Agrees not to participate in another clinical trial at any time during the study period.
* Agrees to remain in the Baltimore-Washington metropolitan area for 7 days after vaccination.

Exclusion Criteria:

* History of any of the following medical illnesses:

  * Toxic shock syndrome
  * Asthma requiring daily prescription medication
  * Psychiatric disorder requiring hospitalization
  * Anaphylaxis/hypersensitivity reactions to glycine, or alum (vaccine components)
  * Coagulopathy
  * Kidney disease
  * Diabetes
  * Cancer
  * Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
  * Vascular disease (peripheral vascular disease, coronary artery disease, stroke)
  * Arthritis
  * Autoimmune disease (e.g., lupus erythematosis, rheumatoid arthritis)
  * Unconsciousness (other than a single brief "concussion")
  * Seizures (other than febrile seizures as a child <5 years old)
  * Recurrent infections (more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
  * Any current illness requiring regular medication therapy other than vitamins or birth control
* Any clinically significant abnormality including but not limited to:

  * Murmur (other than a functional murmur)
  * Focal neurological
  * Hepatosplenomegaly
  * Lymphadenopathy
  * Jaundice
* Lab abnormality, as listed below. Toxicity grading scale provided in Appendix B, Normal ranges provided in Appendix C. Laboratories with abnormalities possibly transient in nature may be repeated one time.

  * Hemoglobin, White blood cell count, Neutrophil count, or Platelet count outside the normal range
  * PT, PTT above the normal range
  * Sodium, or potassium outside the normal range
  * Creatinine above normal range
  * Glucose outside the normal range (65 to <110 mg/dL is acceptable if non-fasting test)
  * AST, ALT, alkaline phosphatase, total bilirubin of grade 1 or greater on the toxicity grading scale
  * Urinalysis with proteinuria or hematuria
  * Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen (Subjects will be informed if their results are positive for hepatitis C, HIV antibody or hepatitis B surface antigen and will be referred to a primary care provider for follow up of these abnormal laboratory tests.)
* Have a positive urine drug screen.
* For women, positive serum pregnancy test within 45 days and urine pregnancy test within 24 hours of administering STEBVax at days 0 and for the highest dose group who receive two doses of vaccine, on day 21.
* Nursing mother
* Temperature > 38.0 degrees C (100.4 degrees F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days before administration of STEBVax
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Failure to pass written examination (70 percent correct answers required to pass) on the first attempt. (The exam is administered to assess and document comprehension of the material presented which covers all aspects of the study including the purpose, procedures, risks, benefits and pertinent microbiology).
* Receipt of an experimental agent (vaccine, drug, device, etc.) within 28 days before administration of STEBVax or expects to receive an experimental agent during the study period.
* Receipt of any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before vaccination in this study or expects to receive a licensed vaccine before vaccination in this study.
* Known sensitivity to any ingredient in STEBVax (recombinant protein, glycine, sodium chloride, alum)
* Prosthetic joint
* Receipt of immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Data describing safety of Staphylococcal Enterotoxin B Vaccine (STEBVax) (clinical observations and clinical laboratory measurements) given in one of several escalating doses. | Through Day 56.

SECONDARY OUTCOMES:
The rate and titer of seroconversion with serum immunoglobulin G (IgG) anti-Staphylococcus aureus enterotoxin B antibodies by enzyme-linked immunosorbent assay (ELISA). | Day 56 and, for the two-dose group, day 77 (56 days after the second dose).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chen WH, Pasetti MF, Adhikari RP, Baughman H, Douglas R, El-Khorazaty J, Greenberg N, Holtsberg FW, Liao GC, Reymann MK, Wang X, Warfield KL, Aman MJ. Safety and Immunogenicity of a Parenterally Administered, Structure-Based Rationally Modified Recombinant Staphylococcal Enterotoxin B Protein Vaccine, STEBVax. Clin Vaccine Immunol. 2016 Dec 5;23(12):918-925. doi: 10.1128/CVI.00399-16. Print 2016 Dec. PMID 27707765